CLINICAL TRIAL: NCT01684865
Title: Prospective, Non Interventional Study to Evaluate the Safety Profile of First- Line Rituximab Maintenance Therapy in Patients With Follicular Non-Hodgkin's Lymphoma
Brief Title: An Observational Study of First-Line Maintenance Rituximab (MabThera/Rituxan) in Participants With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27993
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non-Hodgkin's Lymphoma Participants: Participants initiated on rituximab maintenance therapy according to the standard of care and in line with the current summary of product characteristics will receive rituximab for maximum two years or until disease progression. Participants will be followed for one year after last dose of rituximab administered as maintenance.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Due to observational nature of the study protocol does not specify any dosing schedule for rituximab.
  Other Names: MabThera®, Rituxan®

SUMMARY:
This prospective observational study will evaluate the safety and efficacy of first-line rituximab maintenance therapy in participants with follicular non-Hodgkin's lymphoma. Participants initiated on rituximab maintenance therapy according to the standard of care and in line with the current summary of product characteristics will be followed for a maximum of 3 years or until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of follicular non-Hodgkin's lymphoma
* Complete or partial response to first-line induction therapy with chemotherapy with rituximab
* Participants about to receive first-line rituximab maintenance treatment for follicular non-Hodgkin's lymphoma according to the local label

Exclusion Criteria:

* Pregnant or lactating women
* Receipt of an investigational drug within 30 days prior to initiation of observational drug
* Any medical or psychological alteration that, to criterion of the investigator, can jeopardize the capacity of the participant to grant informed consent
* Central nervous system involvement
* Hepatitis B or C virus infection or human immunodeficiency virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with follicular non-Hodgkin's lymphoma receiving first-line rituximab maintenance treatment
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to approximately 3 years

SECONDARY OUTCOMES:
Progression-Free Survival, as Assessed by Criteria for Evaluation of Response in Non-Hodgkin's Lymphoma | Baseline up to disease progression or death (assessed at baseline and every 8 weeks during 2-year maintenance period and thereafter every 3 months during 1-year follow up period until disease progression or death [up to approximately 3 years])
Time to Progression, as Assessed by Criteria for Evaluation of Response in Non-Hodgkin's Lymphoma | Baseline up to disease progression or death (assessed at baseline and every 8 weeks during 2-year maintenance period and thereafter every 3 months during 1-year follow up period until disease progression or death [up to approximately 3 years])
Time to Next Anti-Lymphoma Treatment (TTNLT) | Baseline up to institution of a new regimen (chemotherapy, radiotherapy or immunotherapy) (up to approximately 3 years)
Time to Next Chemotherapy Treatment (TTNCT) | Baseline up to institution of a chemotherapy regimen or cytotoxic agent or radio-immunotherapy (up to approximately 3 years)
Overall Survival | Baseline up to death (up to approximately 3 years)
Event-Free Survival, as Assessed by Criteria for Evaluation of Response in Non-Hodgkin's Lymphoma | Baseline up to disease progression or death (assessed at baseline and every 8 weeks during 2-year maintenance period and thereafter every 3 months during 1-year follow up period until disease progression or death [up to approximately 3 years])
Percentage of Participants with Overall Response of Complete (CR/CRu) or Partial Response, as Assessed by Criteria for Evaluation of Response in Non-Hodgkin's Lymphoma | Baseline up to disease progression or death (assessed at baseline and every 8 weeks thereafter until disease progression or death [till the end of rituximab maintenance therapy, up to 2 years])

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- University Clinic of Hematology Skopje, Hospital Care Department, Skopje, North Macedonia